CLINICAL TRIAL: NCT00995072
Title: Comparative Effects of Nebivolol and Metoprolol on Female Sexual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Coast Institute for Research (Network)
Responsible Party: Principal Investigator, Benjamin Epstein, Principal Investigator, East Coast Institute for Research
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAIRB-09-0011
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hypertension; Female Sexual Dysfunction
Keywords: sexual dysfunction; female; hypertension; high blood pressure; beta blockers; metoprolol; nebivolol; Bystolic; Toprol XL
MeSH Terms: conditions — Hypertension; Sexual Dysfunction, Physiological | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Nebivolol 5 mg daily for 12 weeks followed by Metoprolol succinate 100 mg daily for 12 weeks. A two week washout (no medication) is completed prior to switching to metoprolol.
  Interventions: Drug: nebivolol and metoprolol succinate
- Arm B (Experimental): Metoprolol succinate 100 mg daily for 12 weeks followed by nebivolol 5 mg daily for 12 weeks. A two week washout (no medication) is completed prior to switching to nebivolol.
  Interventions: Drug: metoprolol succinate and nebivolol

INTERVENTIONS:
Drug: nebivolol and metoprolol succinate — Subjects randomized to treatment Arm A will receive nebivolol 5 mg once daily for 12 weeks. After 12 weeks, double blind therapy will be discontinued and patients will undergo a wash-out period of study therapy over 2 weeks. Subjects randomized to treatment Arm A will then receive metoprolol succinate 100 mg once daily. Subjects will continue double blind therapy for a total duration of 12 weeks.
  Other Names: nebivolol; Bystolic; metoprolol succinate; Toprol XL
  Arms: Arm A
Drug: metoprolol succinate and nebivolol — Subjects randomized to treatment Arm B will receive metoprolol succinate 100mg once daily for 12 weeks. After 12 weeks, double blind therapy will be discontinued and patients will undergo a wash-out period of study therapy over 2 weeks. Subjects randomized to treatment Arm B will then receive nebivolol 5 mg once daily. Subjects will continue double blind therapy for a total duration of 12 weeks.
  Other Names: nebivolol; Bystolic; metoprolol succinate; Toprol XL
  Arms: Arm B

SUMMARY:
Beta-blockers (BB) are an important treatment for high blood pressure and heart disease. However beta-blockers can cause sexual dysfunction (SD) and this common side effect limits successful use of this class of medications. Sexual side effects often result in drug discontinuation, compromising therapy goals. The investigators are conducting the study to determine if nebivolol, a newer beta blocker that is selective for receptors in the heart and causes vasodilation in the body causes fewer sexual side effects, or even improves sexual function, compared with metoprolol succinate.

DETAILED DESCRIPTION:
This protocol is designed to compare the effects two beta blockers, nebivolol (Bystolic) 5-10 mg daily with metoprolol succinate (Toprol XL) 100-200 mg daily on sexual function in post-menopausal women with high blood pressure. The study is composed of 2 treatment phases. At baseline subjects are randomized to either nebivolol 5 mg once daily or metoprolol succinate 100 mg once daily. After randomization, subjects are treated for 12 weeks with double blind therapy. Following double-blind therapy subjects enter a 2-week washout phase and are subsequently switched to the alternate therapy.

After 4 weeks (visits 3 and 7) of double-blind treatment with either nebivolol 5 mg once daily or metoprolol succinate 100 mg once daily subjects will be evaluated and the need for dosage titration assessed. If blood pressure is not at goal the dosage of study medication will be doubled to nebivolol 10 mg once daily or metoprolol succinate 200 mg once daily. If blood pressure remains uncontrolled after 8 weeks of double blind treatment with study medication open label amlodipine 5 mg will be initiated (visits 4 and 8) at the discretion of the principal investigator. During double blind treatment subjects will be evaluated in clinic every 4 weeks.

The primary efficacy variable is the change from baseline in Changes in Sexual Functioning Questionnaire (CSFQ) and the Female Sexual Function Index (FSFI).

The primary study objective is to determine whether nebivolol causes fewer sexual side effects compared with metoprolol succinate and if nebivolol improves FSF in women. FSF will be assessed with the above questionnaires-FSFI and CSFQ.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 40 years
2. Postmenopausal (according to self report of 12 consecutive months of amenorrhea, serum FSH concentrations greater than 40 international units/L, or surgical history consistent with menopause)
3. In a stable monogamous relationship with a male partner for at least 6 months
4. History of hypertension, treated or untreated
5. Requirement for the initiation of an anti-hypertensive agent OR addition of another anti-hypertensive medication (according to the principal investigator and based on clinical judgment) OR patients requiring monotherapy with an anti-hypertensive that wish to participate in the study and are willing to undergo a two week wash-out of current anti-hypertensive therapy
6. Provide written informed consent prior to participation.

Exclusion Criteria:

1. Properly measured clinic SBP > 170 mmHg
2. Advanced AV block
3. Severe hepatic disease
4. Heart rate < 55 beats/min (and not currently on beta blocker therapy)
5. Pregnancy or lactation
6. Heart failure with ejection fraction less than 0.40
7. History of myocardial infarction
8. History of Raynaud's syndrome
9. Patients with alcoholism or recreational drug use will be excluded due to concerns about the ability to comply with the study requirements.
10. Major psychiatric disorder not well controlled with treatment
11. Spinal cord injury
12. Severe respiratory disease, which in the opinion of the investigator contraindicates BB treatment
13. Poorly controlled diabetes mellitus (≥ 9%)
14. Persistent arrhythmia

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Epstein, PharmD, Principal Investigator — East Coast Institute for Research
Locations (1):
- Family Practice, Jacksonville, Florida, United States

REFERENCES:
- See also: Related Info — http://www.eastcoastresearch.net

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 subjects were randomized and dropped from the study prior to taking the study medication
Groups:
- Nebivolol 5 mg Daily First, Then Metoprolol Succinate 100 mg: Nebivolol 5 mg daily for 12 weeks followed by Metoprolol succinate 100 mg daily for 12 weeks. A two week washout (no medication) is completed prior to switching to metoprolol.
  nebivolol and metoprolol succinate: Subjects randomized to treatment Arm A will receive nebivolol 5 mg once daily for 12 weeks. After 12 weeks, double blind therapy will be discontinued and patients will undergo a wash-out period of study therapy over 2 weeks. Subjects randomized to treatment Arm A will then receive metoprolol succinate 100 mg once daily. Subjects will continue double blind therapy for a total duration of 12 weeks.
- Metoprolol Succinate 100 mg First, Then Nebivolol 5 mg Daily: Metoprolol succinate 100 mg daily for 12 weeks followed by nebivolol 5 mg daily for 12 weeks. A two week washout (no medication) is completed prior to switching to nebivolol.
  metoprolol succinate and nebivolol: Subjects randomized to treatment Arm B will receive metoprolol succinate 100mg once daily for 12 weeks. After 12 weeks, double blind therapy will be discontinued and patients will undergo a wash-out period of study therapy over 2 weeks. Subjects randomized to treatment Arm B will then receive nebivolol 5 mg once daily. Subjects will continue double blind therapy for a total duration of 12 weeks.
Period: Overall Study
Arm/Group | Nebivolol 5 mg Daily First, Then Metoprolol Succinate 100 mg | Metoprolol Succinate 100 mg First, Then Nebivolol 5 mg Daily
Started | 10 | 15
Completed | 9 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol 5 mg Daily First, Then Metoprolol Succinate 100 mg | Metoprolol Succinate 100 mg First, Then Nebivolol 5 mg Daily | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Categorical [Count of Participants; unit: Participants] — Population: The number analysed in rows differs from overall due to dropouts.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 8 | 9 | 17
    >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Female Sexual Function Index
Description: This scale is a self-reported instrument used to detect female sexual function. The scale ranges from 2 to 36. The higher score indicates higher sexual function.
Time Frame: Baseline, 12 weeks
Population: The number of participants analyzed for the measure are participants that had data available for both of the study periods.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nebivolol 5 mg Daily: Nebivolol 5 mg daily for 12 weeks
- Metoprolol Succinate 100 mg Daily: Metoprolol succinate 100 mg daily for 12 weeks
Arm/Group | Nebivolol 5 mg Daily | Metoprolol Succinate 100 mg Daily
Number analyzed (Participants) | 15 | 15
units on a scale | 1.24 (9.183) | 1.42 (5.262)

2. Secondary Outcome: Change in Sexual Functioning Questionnaire Score
Description: This scale is a self-reported instrument used to detect sexual functioning. The scale ranges from 14 to 70. The higher scores reflects higher sexual functioning.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebivolol 5 mg Daily | Metoprolol Succinate 100 mg Daily
Number analyzed (Participants) | 13 | 13
units on a scale | 2.38 (7.600) | 0.85 (8.315)

ADVERSE EVENTS:
Description: Adverse Events were collected but the data were destroyed and are not available for reporting.
Groups:
- Nebivolol 5 mg: Nebivolol 5 mg daily
- Metoprolol Succinate 100 mg: Metoprolol succinate 100 mg daily
Arm/Group | Nebivolol 5 mg | Metoprolol Succinate 100 mg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study had a lower than anticipated enrollment and a high drop-out rate due to loss of follow-up-although the drop-out rate was not unexpected based on the study population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No